CLINICAL TRIAL: NCT00501124
Title: Phase IV Study to Evaluate the Safety and Efficacy of Clevudine Compared With Clevudine and Vaccine in Patients Chronically Infected With HBV, HBeAg(+)
Brief Title: Safety and Efficacy Study of Clevudine Compared With Clevudine and Vaccine in Patient With HBeAg(+) Chronic HBV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bukwang Pharmaceutical (Industry)
Responsible Party: HY Lee, Chungnam University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L-FMAU-402
Record Dates: First submitted 2007-07-12; First posted 2007-07-13 (Estimated); Last update posted 2010-12-22 (Estimated); Status verified 2009-08

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — clevudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Clevudine
Biological: Purified hepatitis B surface antigen

SUMMARY:
A randomized, parallel, multicenter, active-controlled with 48 weeks of treatment period. Patients will be randomized to receive clevudine alone for 48 weeks or clevudine for 24 weeks followed by 24 weeks of clevudine in addition to monthly HBV vaccination.The purpose of this study is to investigate efficacy of combination of clevudine and HBV vaccine over clevudine alone in patients with chronic hepatitis B infection.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is between 18 and 60
2. Patient is HBV DNA positive with DNA levels ≥ 5 x 10(6) copies/mL within 30 days of baseline.
3. Patient is documented to be HBsAg positive for > 6 months. Patient is HBeAg positive.
4. Patient has ALT levels which are in the range of ≥2 x ULN/L at least 2 consecutive visits, at least one month apart and bilirubin levels less than 2.0 mg/dL, prothrombin time of less than 1.7 (INR), a serum albumin level of at least 3.5 g/dL.
5. Women of childbearing potential must have a negative urine (β-HCG) pregnancy test taken within 14 days of starting therapy.
6. Patient is able to give written informed consent prior to study start and to comply with the study requirements.

Exclusion Criteria:

1. Patient is currently receiving antiviral, immunomodulatory, cytotoxic or corticosteroid therapy.
2. Patients previously treated with interferon, lamivudine, adefovir, entecavir, telbivudine or any other investigational nucleoside for HBV infection.
3. Patient has a history of ascites, variceal hemorrhage or hepatic encephalopathy.
4. Patient is coinfected with HCV, HDV or HIV.
5. Patient with clinical evidence of decompensated liver disease or HCC
6. ANA > 1:160 and positive anti-smooth muscle antibody as evidence of autoimmune hepatitis
7. Patient is pregnant or breast-feeding.
8. Patient is unwilling to use an "effective" method of contraception during the study and for up to 3 months after the use of study drug ceases.
9. Patient has a clinically relevant history of abuse of alcohol or drugs.
10. Patient has a significant immunocompromised, gastrointestinal, renal, hematological, psychiatric, bronchopulmonary, biliary diseases excluding asymptomatic GB stone, neurological, cardiac, oncologic or allergic disease or medical illness that in the investigator's opinion might interfere with therapy. The patient with a benign tumor, excluded if judged by an investigator that the continuation of study would be interfered by the tumor.
11. Patient has creatinine clearance less than 60mL/min as estimated by the following formula: (140-age in years) (body weight [kg])/(72) (serum creatinine [mg/dL]) [Note: multiply estimates by 0.85 for women]

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2007-05; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Antiviral Activity: Proportion of patients with HBeAg loss | Screening, Day1(predose), every 4 weeks during treatment period(48weeks)
Safety Endpoints:Laboratory tests, Adverse Events, Vital signs, ECG | Screening, Day1(predose), every 4 weeks during treatment period(48weeks), ECG: screening, Week48

SECONDARY OUTCOMES:
Proportion of patients with HBV DNA below LOD, Biochemical improvement, Proportion of patients with seroconversion | Screening, Day1(predose), every 4 weeks during treatment period(48weeks)
Immunological endpoints: Alterations in immunological parameters before, after therapy, particularly with regards to the proliferative a | Day1(predose), Week 8, 16, 24, 28, 32, 40 and 48

CONTACTS AND LOCATIONS:
Overall Officials: Heon Young Lee, MD. PhD., Principal Investigator — Chungnam National University Hospital; Hyeon Woong Yang, MD. PhD., Principal Investigator — Eulji University Hospital
Locations (7):
- South Korea (7):
  - Dankook University Hospital, Anseo-dong, Cheonan Si, Chungcheongnam-do
  - Soon Chun Hyang University Cheonan Hospital, Bongmyeong-dong, Cheonan Si, Chungcheongnam-do
  - The Catholic University of Korea, Daejeon St. Mary's Hospital, Daeheung-dong, Jung-gu, Daejeon
  - Chungnam National University Hospital, Daesa-dong, Jung-gu, Daejeon
  - Eulji University Hospital, Dunsan 2-dong, Seo-gu, Daejeon
  - Konyang University Hospital, Gasuwon-dong, Seo-gu,, Daejeon
  - Chungbuk National University Hospital, Gaesin-dong, Cheongju Si Heungdeok-gu, North Chungcheong